CLINICAL TRIAL: NCT02762526
Title: Repercussions of Lipoabdominoplasty Surgery on Diaphragmatic Mobility, Regional Distribution Ventilation of Thoracoabdominal System and Lung Function in Women Healthy.
Brief Title: Lipoabdominoplasty and Diaphragmatic Mobility
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Sandra Fluhr Souto Barros, MASTER STUDENT, Universidade Federal de Pernambuco
Other Study IDs: SF-6671649
Record Dates: First submitted 2016-04-27; First posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Abdominoplasty Surgery
Keywords: lipectomy; abdominoplasty; plethysmography optoelectronics; diaphragmatic mobility; lung function; respiratory muscles
MeSH Terms: interventions — Lipoabdominoplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Lipoabdominoplasty

SUMMARY:
Background: The lipoabdominoplasty can lead to respiratory complications in the postoperative period becoming critical early clinical and functional evaluation of respiratory muscles, seeking to direct a more effective treatment, which can result in shorter hospital stays and lower spending on health in patients undergoing such procedures. Objective: To evaluate the correlation of regional distribution of ventilation system with thoracoabdominal diaphragmatic mobility in women undergoing surgery lipoabdominoplasty comparing preoperative, 10 ° and 30 ° DPO DPO. Methods: This is a prospective cohort study, which will be evaluated 30 women aged 25 to 55 years undergoing lipoabdominoplasty surgery without respiratory or prior cardiac comorbidities and body mass index (BMI) ≤ 30 kg / cm2. women smokers are deleted and / or a history of smoking more than 10 years and unable to understand the commands to perform the proposed methods. For evaluation of diaphragmatic mobility will be used high-resolution ultrasound with convex 3.5 MHz transducer. The evaluation of the regional distribution of ventilation thoracoabdominal system will be made using the optoelectronic plethysmograph (POE). The strength of the inspiratory and expiratory muscles is measured through a digital manometer connected to a nozzle with an orifice of 2 mm to reduce the closing pressure of the glottis. A portable spirometer is used for assessment of pulmonary function and evaluation of dyspnea will be used modified Borg scale. The data will be evaluated in the preoperative period, 10 days and 30 days postoperatively. Hypotheses: Patients undergoing surgery lipoabdominoplasty have decreased diaphragmatic mobility, strength and respiratory function, in addition to presenting changes in the pattern of regional ventilation distribution in torocoabdominal system in the postoperative period when compared to the preconditions surgery.

DETAILED DESCRIPTION:
Introduction:

The lipoabdominoplasty can lead to respiratory complications in the postoperative period becoming critical early clinical and functional evaluation of respiratory muscles, seeking to direct a more effective treatment, which can result in shorter hospital stays and lower spending on health in patients subjected to this type of procedure.

hypotheses: Patients undergoing lipoabdominoplasty surgery with muscular plication, have decreased diaphragmatic mobility, strength and respiratory function, in addition to presenting changes in the regional distribution pattern of ventilation in torocoabdominal system in the postoperative period when compared to the preconditions surgery .

Goal:

To evaluate the correlation of regional distribution of ventilation system with thoracoabdominal diaphragmatic mobility in women undergoing surgery lipoabdominoplasty comparing preoperative, 10 ° and 30 ° DPO DPO.

Hypothesis:

Patients undergoing surgery lipoabdominoplasty have decreased diaphragmatic mobility, strength and respiratory function, in addition to presenting changes in the pattern of regional ventilation distribution in torocoabdominal system in the postoperative period when compared to the preconditions surgery.

Materials and methods:

This is a prospective cohort study, which will be evaluated 30 women between 30 and 50 years underwent surgery lipoabdominoplasty without respiratory or prior cardiac comorbidities and body mass index (BMI) ≤ 30 kg / cm2. women smokers are deleted and / or a history of smoking greater than 10 years, FEV1 <80% predicted, FEV1 / FVC <70% of predicted and unable to understand the commands to perform the proposed methods. For evaluation of diaphragmatic mobility and thickness will be used high-resolution ultrasound with a convex transducer of 3.5 MHz and 7.5 MHz linear transducer, respectively. The assessment of the regional distribution of ventilation thoracoabdominal system will be made using the optoelectronic plethysmograph (POE). The strength of the inspiratory and expiratory muscles is measured through a digital manometer connected to a nozzle with an orifice of 2 mm to reduce the closing pressure of the glottis. A portable spirometer is used for assessment of pulmonary function and evaluation of dyspnea will be used modified Borg scale. The data will be evaluated in the preoperative period, 10 days and 30 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* women will be included between 25 and 55 years underwent surgery lipoabdominoplasty without respiratory or prior cardiac comorbidities and body mass index (BMI) ≤ 30 kg / cm2.

Exclusion Criteria:

* women smokers will be deleted and / or a history of smoking more than 10 years; FEV1 <80% predicted and FEV1 / FVC <70% of predicted; unable to understand the commands to perform the proposed methods.

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women undergoing lipoabdominoplasty who meet the eligibility criteria for the search.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Mobility Diaphragmatic | 30 days
  Measure diaphragmatic mobility for total lung capacity maneuver
plethysmography optoelectronics | 30 days
  measuring the change in lung volumes in the three compartments

CONTACTS AND LOCATIONS:
Overall Officials: Daniella Araújo, PHD, Study Chair — UFPE

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pereira N, Sciaraffia C, Danilla S, Parada F, Asfora C, Moral C. Effects of Abdominoplasty on Intra-Abdominal Pressure and Pulmonary Function. Aesthet Surg J. 2016 Jun;36(6):697-702. doi: 10.1093/asj/sjv273. Epub 2016 Feb 9. PMID 26895955
- [Result] Rodrigues MA, Nahas FX, Gomes HC, Ferreira LM. Ventilatory function and intra-abdominal pressure in patients who underwent abdominoplasty with plication of the external oblique aponeurosis. Aesthetic Plast Surg. 2013 Oct;37(5):993-9. doi: 10.1007/s00266-013-0158-5. Epub 2013 Aug 27. PMID 23982698
- [Result] Staalesen T, Elander A, Strandell A, Bergh C. A systematic review of outcomes of abdominoplasty. J Plast Surg Hand Surg. 2012 Sep;46(3-4):139-44. doi: 10.3109/2000656X.2012.683794. Epub 2012 Jul 2. PMID 22747350
- [Result] Tercan M, Bekerecioglu M, Dikensoy O, Kocoglu H, Atik B, Isik D, Tercan A. Effects of abdominoplasty on respiratory functions: a prospective study. Ann Plast Surg. 2002 Dec;49(6):617-20. doi: 10.1097/00000637-200212000-00011. PMID 12461445
- [Result] Perin LF, Saad R Jr, Stirbulov R, Helene A Jr. Spirometric evaluation in individuals undergoing abdominoplasty. J Plast Reconstr Aesthet Surg. 2008 Nov;61(11):1392-4. doi: 10.1016/j.bjps.2008.02.028. Epub 2008 Aug 8. No abstract available. PMID 18693147
- [Derived] Fluhr S, Andrade AD, Oliveira EJB, Rocha T, Medeiros AIC, Couto A, Maia JN, Brandao DC. Lipoabdominoplasty: repercussions for diaphragmatic mobility and lung function in healthy women. J Bras Pneumol. 2019 May 30;45(3):e20170395. doi: 10.1590/1806-3713/e20170395. PMID 31166554
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed